CLINICAL TRIAL: NCT04182347
Title: Engagement in Healthy Communities for People With Intellectual and Developmental Disabilities
Brief Title: Research Engagement With People With Intellectual and Developmental Disabilities
Acronym: PCORI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018-1215; A176000 (Other: UW Madison); EDUC/KINESIOLOGY (Other: UW Madison)
Record Dates: First submitted 2019-10-22; First posted 2019-12-02 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Intellectual Disability; Developmental Disability; Chronic Conditions, Multiple
Keywords: Individuals with Intellectual or Developmental Disabilities; Research; ToolKit; Health Disparities; Engagement
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities; Multiple Chronic Conditions

STUDY DESIGN:
Intervention Model Description: A ToolKit will be created to support the engagement of people with IDD in the development of research. The toolkit will be the first of its kind to provide an accessible, structured process with the necessary training for people with IDD and people with IDD's paid and unpaid caregivers to be engaged partners. Learning activities are focused on leadership, information about research, health for individuals with IDD. Learning activities will include topics:
  What is health research? What is the health research process? How can individuals with IDD be involved in health research? Where is research happening? How to think like a researcher. Creating health stories for research and care advocacy.
  The learning activities will teach individuals with IDD information and allow participants to practice the learning.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People with IDD and caregivers (Other)
  Interventions: Other: Health Research ToolKit Development

INTERVENTIONS:
Other: Health Research ToolKit Development — The Toolkit will be an accessible, structured process for people with IDD and people with IDD's paid and unpaid caregivers to be engaged partners. Learning activities are focused on leadership, information about research, health for individuals with IDD. Learning activities will include topics:
  What is health research? What is the health research process? How can individuals with IDD be involved in health research? Where is research happening? How to think like a researcher. Creating health stories for research and care advocacy.
  The learning activities will teach individuals with IDD information and allow participants to practice the learning.
  Other Names: Learning Activities

SUMMARY:
The objectives of this project are to to build sustainable regional communities of Intellectual or Developmental Disabilities (IDD) stakeholders to provide ongoing input to research priorities, methodological processes, and relevant person-centered health outcomes; leverage existing Special Olympic infrastructure to nationally disseminate the toolkit in order to increase participation and engagement in research and improve health outcomes; conduct comparative effectiveness trials that incorporate people with IDD focusing on their research priorities.

DETAILED DESCRIPTION:
This project will develop a skilled community of stakeholders through collaboration with Special Olympics to create capacity building working groups. Groups will collaborate to develop stakeholder training modules focused on leadership, research fundamentals, and health. Collaboratively developed trainings will be piloted to support revising of the Toolkit for the engagement of people with IDD in research. A range of stakeholders will be essential members of the team to design and provide critical feedback on the effectiveness of the Toolkit, research priorities, and ecologically valid methodologies. Finally, research priorities will be refined, and the research engagement Toolkit will be nationally disseminated to Special Olympics and relevant community organizations. The toolkit will include necessary training for people with IDD, as well as paid and unpaid caregivers to be engaged partners in research.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Intellectual or Developmental Disabilities (IDD)
* Caregiver or family member of the individual with IDD
* Patients/consumer
* Clinician
* Complete informed consent or assent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
READI Curriculum Development | Up to one year
  The development of an online health research curriculum incorporating stakeholders as part of the development team.
Health Research Infographic Development | Up to one year
  The development of health research infographics incorporating stakeholders as part of the development team that will bridge knowledge dissemination between researchers and people with IDD.

CONTACTS AND LOCATIONS:
Locations (1):
- Waisman Center, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No